CLINICAL TRIAL: NCT00250250
Title: An Open-Label, Multi-centre, Phase III Study of Local Tolerability of ZOMACTON 10MG (Recombinant Somatropin) Administered by ZomaJet Vision X
Brief Title: An Open-Label, Multi-centre, Phase III Study of Local Tolerability of ZOMACTON 10MG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE999905 CS002
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Turner's Syndrome
MeSH Terms: conditions — Turner Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ZOMACTON

SUMMARY:
Children with growth failure due to inadequate secretion of growth hormone or growth retardation due to Turner's syndrome are individually dosed and treated for 12 weeks

DETAILED DESCRIPTION:
Ferring Pharmaceuticals A/S has developed a new ZOMACTON 10 mg formulation. The formulation provides a higher concentration and thereby a smaller volume to be administered. ZomaJet Vision X is a needle-free injection system. It sends a thin jet of ZOMACTON through the skin and into the subcutaneous tissue without the use of a needle. The mode of administration is referred to as "transjection". By use of ZomaJet Vision X, both transjection and reconstitution of ZOMACTON 10 mg can be done without using a needle. The rationale of the study is to describe the local tolerability of the new ZOMACTON 10 mg administered by ZomaJet Vision X.

ELIGIBILITY:
Subjects between the ages of 3 and 17 years (both inclusive) with growth failure due to inadequate secretion of growth hormone or growth retardation due to Turner's syndrome. Subjects have for a minimum of 6 months prior to study enrolment been receiving growth hormone therapy

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To assess the local tolerability of an individualised dose of ZOMACTON 10 mg administered by ZomaJet Vision X

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (6):
- Czechia (3):
  - Faculty Hospital Olomouc, Children's Clinic, Endocrinology Outpatient Department, I.P.Pavlova str. 6,, Olomouc
  - Faculty Hospital Kralovske Vinohrady, Children's Clinic, Vinohradska str. 159, Prague
  - Masaryk Hospital Usti nad Labem, Children's Clinic, Building D2, Endocrinology Outpatient Department, Socialni pece 12a, Ústí nad Labem
- France (2):
  - Centre d'Endocrinologie Pediatrique, 25 rue Boudet, Bordeaux
  - Service de Pédiatrie, Groupe Hospitalier du Havre, 55 bis, rue Gustave Flaubert, Le Havre
- Vu medisch centrum, Paediatrics, De Boelelaan 1117, PO Box 7057, Amsterdam, Netherlands